CLINICAL TRIAL: NCT06981442
Title: Implementation and Evaluation of Vector Control Methods in Kinshasa: The Case of Aedes, Vectors of Arboviruses.
Brief Title: Implementation and Evaluation of Vector Control Methods in Kinshasa: The Case of Aedes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National de Recherche Biomédicale. Kinshasa, République Démocratique du Congo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1778/24
Record Dates: First submitted 2025-04-08; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Aedes-borne Diseases
Keywords: Vector control; Aedes mosquitoes; Democratic Republic of the Congo
MeSH Terms: conditions — Mosquito-Borne Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ARM 1_Community-based environmental management (Experimental): This intervention will be carried out by the community, who will have received training and information on the environmental management measures suitable for controlling the Aedes mosquito. It will involve a cluster of 400 households randomly assigned to this intervention.
  Interventions: Behavioral: Community-based environmental management
- ARM 2_Community-based environmental management AND vector control against immature stages of Aedes (Experimental): This intervention combines community-based environmental management (specified in the first study arm) with vector control against immature stages of Aedes. It will involve a cluster of 400 households randomly assigned to this intervention.
  Interventions: Behavioral: Community-based environmental management; Other: Vector control against immature stages of Aedes
- ARM 3_Community-based environmental management AND vector control against mature stages of Aedes (Experimental): This intervention combines community-based environmental management (specified in the first arm of the study) with vector control against the mature stages of Aedes. It will involve a cluster of 400 households randomly assigned to this intervention.
  Interventions: Behavioral: Community-based environmental management; Other: Vector control against the mature stages of Aedes
- ARM 4_Control arm (No Intervention): No control interventions will be implemented. It will involve a cluster of 400 households randomly assigned to this arm.

INTERVENTIONS:
Behavioral: Community-based environmental management — This intervention will be performed by the local community, who will have been previously informed and trained on the appropriate environmental management methods for the control of the Aedes mosquito. It will be based on the following elements: i) identification and removal of all artificial sources of reproduction of the Aedes mosquito inside and around the house (i.e. covering abandoned containers and/or storage containers to avoid water accumulation); ii) regular collection and disposal of household waste; iii) identification and resolution of all artificial sources of reproduction of the Aedes vector in or around the house (i.e. natural cavities such as tree holes will be filled to prevent water accumulation). This intervention will be carried out as a single intervention in Arm 1, in combination with a larvicidal intervention in Arm 2 and in combination with the intervention against the adult stage of the Aedes mosquito in Arm 3.
  Arms: ARM 1_Community-based environmental management; ARM 2_Community-based environmental management AND vector control against immature stages of Aedes; ARM 3_Community-based environmental management AND vector control against mature stages of Aedes
Other: Vector control against immature stages of Aedes — Larvicidal control will be carried out through pyriproxifen-based autodissemination stations combined with Beauveria bassiana, implemented according to the manufacturer's recommended procedures.
  Arms: ARM 2_Community-based environmental management AND vector control against immature stages of Aedes
Other: Vector control against the mature stages of Aedes — The control of the adult Aedes mosquitoes will be carried out through mass trapping using BG-GAT traps implemented according to the manufacturer's recommended procedures. In each household, three traps will be deployed.
  Arms: ARM 3_Community-based environmental management AND vector control against mature stages of Aedes

SUMMARY:
Arboviral diseases are viral diseases transmitted by mosquitoes of the Aedes genus and are constantly spreading throughout the world, constituting a significant threat to public health.

In Africa, there is very little data on the epidemiological situation of Aedes-borne diseases and programs for monitoring these diseases are very limited. In the Democratic Republic of the Congo (DRC), several epidemics of yellow fever, dengue fever, chikungunya and Zika cases have been reported. In particular, in Kinshasa, the dengue and chikungunya viruses have previously been detected in patients with undifferentiated fevers and several studies have shown entomological transmission indices above the criteria and standards of the World Health Organization (WHO).

The aim of our study is to implement and evaluate different strategies to control Aedes mosquitoes at different stages of their life cycle in the city of Kinshasa.

In particular, a before-and-after interventional study will be piloted and tested in the health zone of Kinshasa, with the aim of providing preliminary evidence of the impact of vector control tools.

Interventions will be implemented in 400 households for each arm for 12 months. Before, after and during the interventions, entomological surveys will be conducted in 160 households in each arm to define the density of the vectors. Mosquitoes will be tested for the possible presence of arbovirus RNA (dengue, chikungunya, Zika, yellow fever). During the pre-intervention period, a serological survey for the same diseases transmitted by the Aedes mosquito will be conducted on a sample of 450 people included in two health centers of reference for the health zone of Mont Ngafula 1. A questionnaire will also be administered before and after the intervention implementation to assess the community's knowledge, attitudes and practices towards Aedes mosquito vector control and Aedes-borne diseases.

The integration of the data collected within the scope of this study will provide an assessment of the feasibility and impact of the tested methods on entomological indicators, as well as determining the exposure and knowledge of Aedes-borne diseases in the Mont Ngafula 1 area.

DETAILED DESCRIPTION:
Arboviral diseases are viral diseases transmitted by mosquitoes of the Aedes genus and are constantly spreading throughout the world, constituting a significant threat to public health. In the last 30 years, the frequency and extent of Aedes-borne epidemics have increased significantly and the main vectors, Aedes aegypti and Aedes albopictus, have expanded their geographical distribution worldwide.

In Africa, there is very little data on the epidemiological situation of Aedes-borne diseases and programs for monitoring these diseases are very limited. In the Democratic Republic of the Congo (DRC), several epidemics of yellow fever, dengue fever, chikungunya and Zika cases have been reported. In particular, in Kinshasa, the dengue and chikungunya viruses have previously been detected in patients with undifferentiated fevers and several studies have shown entomological transmission indices above the criteria and standards of the World Health Organization (WHO). However, vector control activities for Aedes are not carried out regularly outside of epidemic periods and the need for targeted strategies remains essential.

The aim of our study is to implement and evaluate different strategies to control Aedes mosquitoes at different stages of their life cycle in the city of Kinshasa. Furthermore, the integration of a serological survey on diseases transmitted by the Aedes vector will strengthen our knowledge on the circulation of these diseases in the area, for which the data in the literature remain fragmentary until now.

In particular, a before-and-after interventional study will be piloted and tested in the health zone of Mont Ngafula 1, Kinshasa, which is characterized by ecological diversity and a known history of arbovirus circulation. In this pilot study, with the aim of providing preliminary evidence of the impact of vector control tools, there are four arms: i) community-based environmental management approach, ii) community-based environmental management and vector control against immature stages of Aedes (pyriproxifen-based autodissemination stations), iii) community-based environmental management and vector control against the mature stages of Aedes aegypti (mass trapping using BG-GAT - Gravid Aedes Traps), iv) control arm without implementation of vector control interventions. These interventions will be implemented in 400 households for each arm for 12 months. Before, after and during the interventions, entomological surveys will be conducted in 160 households in each arm to define the density of the vectors. Mosquitoes will be tested for the possible presence of arbovirus RNA (dengue, chikungunya, Zika, yellow fever). During the pre-intervention period, a serological survey for the same diseases transmitted by the Aedes mosquito will be conducted on a sample of 450 people included in two health centers of reference for the health zone of Mont Ngafula 1. The knowledge, attitudes and practices of the subjects belonging to the households enrolled in the study will be collected using an electronic questionnaire before and after the intervention. The integration of the data collected within the scope of this study will provide an assessment of the feasibility and impact of the tested methods on entomological indicators, as well as determining the exposure and knowledge of Aedes-borne diseases in the Mont Ngafula 1 area, for a better definition of the next measures to be adopted in the fight against vectors, tailored to the specific context of the the DRC.

ELIGIBILITY:
At household level:

Inclusion Criteria:

* Belong to a household in one of the 4 health areas selected as study arms
* From 18 years of age to consent for household enrollment and participation in the serosurvey
* Consenting

Exclusion Criteria:

* Not belong to a household in one of the 4 health areas selected as study arms
* Under 18 years of age
* Non-consenting

At health facility level:

Inclusion Criteria:

* From 18 years of age
* Resident of the health zone of Mont Ngafula 1
* Consenting

Exclusion Criteria:

* Under 18 years of age
* Not resident in the health zone of Mont Ngafula 1
* Seriously ill and hospitalized, requiring transfusion, presence of blood clotting disorders, allergies resulting from injections, adverse events associated with previous blood sampling, pregnancy
* Non-consenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2050 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Adult mosquito collection - Entomological Indicator | Six collections in total: 1 at baseline, 4 during the intervention (one per trimester), 1 three months after completion of the intervention.
  Adult mosquitoes will be collected outdoor using Prokopack mosquito aspirator in 50 households at the center of each of the 4 study arms and using BG-Sentinel traps in 10 households at the center of each of the 4 study arms. Adult mosquitoes obtained through BG-GAT traps in Arm 3 will also be collected.
Mosquito larval survey - Entomological Indicator | Six collections in total: 1 at baseline, 4 during the intervention (one per trimester), 1 three months after completion of the intervention.
  Larval surveys will be carried out in 100 households at the center of each of the 4 study arms. Immature mosquitoes obtained through the auto-dissemination stations in Arm 2 will also be collected.
Epidemiological indicator | Once : before/at beginning of intervention
  A sero-survey prospectively including 450 consenting subjects will be carried out in two hospitals in the health zone of Mont Ngafula 1, Kinshasa. The blood sample will be tested for antibodies against the main arboviruses (Yellow Fever, Dengue, Chikungunya, Zika). De-identified socio-demographic data will be collected.

SECONDARY OUTCOMES:
Knowledge, attitudes, and practices. | Twice in total: at the beginning of the study and three months after completion of the intervention.
  A survey on knowledge, practices and behaviors regarding Aedes-borne diseases, Aedes mosquitoes and vector control will be proposed to 100 subjects for each study arm, for a total of 400 participants.

CONTACTS AND LOCATIONS:
Overall Officials: Veerle Vanlerberghe, Principal Investigator — Institute of Tropical Medicine Antwerp
Locations (1):
- Institut National de Recherche Biomédicale, INRB, Kinshasa, République Démocratique Du Congo, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mbanzulu KM, Wumba R, Mukendi JK, Zanga JK, Shija F, Bobanga TL, Aloni MN, Misinzo G. Mosquito-borne viruses circulating in Kinshasa, Democratic Republic of the Congo. Int J Infect Dis. 2017 Apr;57:32-37. doi: 10.1016/j.ijid.2017.01.016. Epub 2017 Jan 30. PMID 28153792
- [Background] Proesmans S, Katshongo F, Milambu J, Fungula B, Muhindo Mavoko H, Ahuka-Mundeke S, Inocencio da Luz R, Van Esbroeck M, Arien KK, Cnops L, De Smet B, Lutumba P, Van Geertruyden JP, Vanlerberghe V. Dengue and chikungunya among outpatients with acute undifferentiated fever in Kinshasa, Democratic Republic of Congo: A cross-sectional study. PLoS Negl Trop Dis. 2019 Sep 5;13(9):e0007047. doi: 10.1371/journal.pntd.0007047. eCollection 2019 Sep. PMID 31487279
- [Background] Selhorst P, Makiala-Mandanda S, De Smet B, Marien J, Anthony C, Binene-Mbuka G, De Weggheleire A, Ilombe G, Kinganda-Lusamaki E, Pukuta-Simbu E, Lubula L, Mbala-Kingebeni P, Nkuba-Ndaye A, Vogt F, Watsenga F, Van Bortel W, Vanlerberghe V, Arien KK, Ahuka-Mundeke S. Molecular characterization of chikungunya virus during the 2019 outbreak in the Democratic Republic of the Congo. Emerg Microbes Infect. 2020 Dec;9(1):1912-1918. doi: 10.1080/22221751.2020.1810135. PMID 32787529
- [Background] Willcox AC, Collins MH, Jadi R, Keeler C, Parr JB, Mumba D, Kashamuka M, Tshefu A, de Silva AM, Meshnick SR. Seroepidemiology of Dengue, Zika, and Yellow Fever Viruses among Children in the Democratic Republic of the Congo. Am J Trop Med Hyg. 2018 Sep;99(3):756-763. doi: 10.4269/ajtmh.18-0156. Epub 2018 Jul 5. PMID 29988000
- [Background] Weetman D, Kamgang B, Badolo A, Moyes CL, Shearer FM, Coulibaly M, Pinto J, Lambrechts L, McCall PJ. Aedes Mosquitoes and Aedes-Borne Arboviruses in Africa: Current and Future Threats. Int J Environ Res Public Health. 2018 Jan 28;15(2):220. doi: 10.3390/ijerph15020220. PMID 29382107